CLINICAL TRIAL: NCT01353495
Title: A Prospective, Randomized Comparative Parallel Study of Acellular Porcine Dermal Matrix Wound Dressing in the Management of Diabetic Foot Ulcers
Brief Title: Acellular Porcine Dermal Matrix Wound Dressing in the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009-BIO-001
Record Dates: First submitted 2011-05-11; First posted 2011-05-13 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APM Graft (BIOTAPE XMTM (Experimental): graft applied to wound q 3 weeks for 12 weeks
  Interventions: Device: APM Graft (BIOTAPE XMTM); Other: Wound Debridement
- standard wound care (Active Comparator): Wound debridement and gels and foams applied to wound weekly for 12 weeks.
  Interventions: Other: Wound Debridement

INTERVENTIONS:
Device: APM Graft (BIOTAPE XMTM) — Patients randomized to the APM group will, following surgical debridement for their diabetic foot wounds, receive a single application of an APM graft (BIOTAPE XMTM, Wright Medical Technology, USA) with dressing changes taking place weekly. All necrotic tissue will be removed from the wound prior to application. BIOTAPE XMTM will be sutured or stapled in place under a silver-based non-adherent dressing (Silverlon, Argenta Medical). Therapy will then be followed by a moisture-retentive dressing (hydrogel bolster) until complete epithelialization has occurred.
  Other Names: BIOTAPE XMTM
  Arms: APM Graft (BIOTAPE XMTM
Other: Wound Debridement — Wounds debrided in both arms of study

SUMMARY:
Have indolent diabetic ulcers completely healed by the Acellular Porcine Dermal Matrix (APM) in 12 weeks.

DETAILED DESCRIPTION:
The primary objective of this study is time -to - healing with wound size determination at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria and Population:

* Male or female age 18 or older
* Informed consent must be obtained
* Patient's ulcer must be diabetic in origin and larger than 1cm2. Debridement will be done prior to randomization. Subject's informed consent for participating in this study, must be obtained prior to proceeding with sharp debridement.
* Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
* Patient's ulcer must exhibit no clinical signs of infection.
* Patient is of legal consenting age.
* Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study.
* Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

  * Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg, OR
  * ABIs with results of ≥0.7 and ≤1.2, OR
  * Doppler arterial waveforms,which are triphasicor biphasic at the ankle of affected leg

Exclusion Criteria:

* Patients presenting with an ulcer probing to bone (UT Grade IIIA-D). A positive probe-to-bone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
* Patients whose index diabetic foot ulcers are greater than 25cm2.
* Patients considered not in reasonable metabolic control, confirmed by an HgA1c greater than 12% within previous 90 days,
* Patients whose serum creatinine levels are 3.0mg/dl or greater.
* Patients with a known history of poor compliance with medical treatments.
* Patients who have been previously randomized into this study, or are presently participating in another clinical trial
* Patients who are currently receiving radiation therapy or chemotherapy.
* Patients with known or suspected local skin malignancy to the index diabetic ulcer.
* Patients on anticoagulant medication will as in any surgical procedure, be monitored According to the protocols employed at the enrolling center.
* Patients diagnosed with autoimmune connective tissues diseases.
* Nonrevascularable surgical sites
* Active infection at site
* Sensitivity to the following antibiotics: Gentamicin, Cefoxilin, Linocmycin, Polymyxin B, Vancomycin
* Any pathology that would limit the blood supply and compromise healing;
* Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagpreet Mukker, DPM, Principal Investigator — Advanced Foot Care and Clinincal Research Center
Locations (2):
- United States (2):
  - Advanced Foot Care and Clinincal Research Center, Fresno, California
  - Professional Education & Research Institute, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects with diabetic wound ulcers were recruited for this study in podiatric wound clinic offices for treatment with the graft or standard wound care. Dates of first enrolled subject was 2010
Pre-assignment Details: an ulcer (UT Grade IIIA-D) index ulcers > than 25cm2 an HgA1c > 12% within previous 90 days, serum cr 3.0mg/dl known history non-compliance previously into this study, or are in another trial receiving radiation therapy,chemotherapy. known local skin malignancy to the index diabetic ulcer. on anticoagulant medication
Groups:
- Standard Wound Care: Standard Wound care (gels, foams, dressings.)
  Wound Debridement : Wounds debrided in both arms of study
- Treatment With Study Device: Treatment with Biotape Acelular Dermis Graft
  APM Graft (BIOTAPE XMTM) : Patients randomized to the APM group will, following surgical debridement for their diabetic foot wounds, receive a single application of an APM graft (BIOTAPE XMTM, Wright Medical Technology, USA) with dressing changes taking place weekly. All necrotic tissue will be removed from the wound prior to application. BIOTAPE XMTM will be sutured or stapled in place under a silver-based non-adherent dressing (Silverlon, Argenta Medical). Therapy will then be followed by a moisture-retentive dressing (hydrogel bolster) until complete epithelialization has occurred.
  Wound Debridement : Wounds debrided in both arms of study
Period: Overall Study
Arm/Group | Standard Wound Care | Treatment With Study Device
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Wound Care | Treatment With Study Device | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 10 | 15 | 25
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Size of Index Wound Based on Calculations Wound Width x Length x Depth 2. Size of Index Wound Based on Calculations Wound Width x Length x Depth
Description: Wound evaluated and granulation described by wound tracing and photographs which will be measures in wound width x length x depth at each week for 12 weeks or until full granulation has occurred in addition to the size of the wound
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Treatment With Study Device | Standard Wound Care
Number analyzed (Participants) | 20 | 19
mm^3 | 2.05 (NA) — data not available as the PI left the institution. Every attempt was made to locate the data, | 3.33 (NA) — data not available as the PI left the institution. Every attempt was made to locate the data,

ADVERSE EVENTS:
Arm/Group | Standard Wound Care | Treatment With Study Device
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 4/19 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Wound Care (N=19) | Treatment With Study Device (N=20)
LT HEEL PAIN WITH POSSIBLE ABSCCESS (Infections and infestations) | 0 (0) | 1 (1) — DEVELOPING PAIN LEFT HEEL OVER PAST FEW DAys; MILD FOWL ODOR &TENDERNESS. ? INFECTION IN THE HEEL. Reported as possibly related to procedure Final report was resolved
RT FOOT INFECTION WITH OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1) — TO HOSPITAL. CELLULITIS RT LEG, FOOT, WAS PLACED ON IV ABX, BONE SCAN ; POSITIVE OSTEOMYELITIS. Reported as possibly related to procedure final eport: resolved reported as possibly related to the device; then reported as resolved
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — PT STARTED EXPERIENCING INCREASING SOB AND COUGHING AND DECIDED TO GO TO ER TO ENSURE NOTHING WAS WRONG. Not related to the device or the procedure Outcome Resolved
CELLULITIS TO THE RIGHT FOOT. (Infections and infestations) | 1 (1) | 0 (0) — SUBJECT HAVING FEVER, CHILLES, AND PAIN. Reported: not related to device or procedure final report: resolved
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 0 (0) — SUBJECT FELL ILL DUE TO FOOD POISONING AND WAS ADMITTED FOR DEHYDRATION OVER THE WEEKEND. reported as unrelated to device or procedure Outcome: resolved
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — SUBJECT WAS HAVING PROBLEM BREATHING Reported as mild Reported as unrelated to device or procedure Reported as Ongoing at the end of the study
DEHYDRATION (Gastrointestinal disorders) | 0 (0) | 1 (1) — SUBJECT FELL ILL DUE TO FOOD POISONING ADMITTED FOR DEHYDRATION OVER THE WEEKEND. Reported as not related to device or procedure final outcome resolved. One foot standard of care other Biotape used

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No